CLINICAL TRIAL: NCT01912833
Title: Assessing the Association Between Stressful Life Events, Hormonal Dysregulation, and Postpartum Depression Among Lactating Latina Mothers: A Pilot Study
Brief Title: Study of Exposure to Stress, Postpartum Mood, Adverse Life Events, and Hormonal Function Among Latinas (SEPAH Latina)
Acronym: SEPAH
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Sandraluz Lara-Cinisomo, PhD, Postdoctoral Fellow, University of North Carolina, Chapel Hill
Other Study IDs: 13-0788
Record Dates: First submitted 2013-07-24; First posted 2013-07-31 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Postpartum Depression
Keywords: postpartum depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oxytocin, cortisol, and adrenocorticotropic hormone (ACTH)

SUMMARY:
The purpose of the funded study is to determine a) examine associations among OT levels, stress, trauma history, PPD, and lactation failure in the full 60-subject sample and assess whether there are differences between immigrant women and non-immigrant Latina women on these measures; b) quantify whether there is a correlation between ACTH, cortisol, and PPD and whether there are differences between immigrant and non-immigrant Latina women; and c) assess the feasibility of enrolling Latinas into a laboratory-based study that includes the collection of venous blood for measurement of oxytocin, ACTH, and cortisol. Sixty prenatal (34 to 37 weeks) Latinas (30 immigrants and 30 U.S.-born) who are between the ages of 18 and 45 will be enrolled. Women with a singleton pregnancy who are Latina, who intend to breastfeed for more than 2 months, who have or do not have a history of depression, and who are willing to be followed for 8 weeks after delivery will be enrolled in the study. Latinas who report maternal or infant disorder that may interfere with breastfeeding; those who endorse substance use, and/or who have or have had a psychiatric disorder (e.g., psychosis or serious personality disorders) other than depression or anxiety will be excluded to minimize risk and confounds with the outcomes of interest.

DETAILED DESCRIPTION:
Study Objective: The purpose of the funded study is to determine a) examine associations among OT levels, stress, trauma history, PPD, and lactation failure in the full 60-subject sample and assess whether there are differences between immigrant women and non-immigrant Latina women on these measures; b) quantify whether there is a correlation between ACTH, cortisol, and PPD and whether there are differences between immigrant and non-immigrant Latina women; and c) assess the feasibility of enrolling Latinas into a laboratory-based study that includes the collection of venous blood for measurement of oxytocin, ACTH, and cortisol.

Research Aims: 1) To examine associations among OT levels, stress, trauma history, PPD, and lactation failure in the full 60-subject sample and assess whether there are differences between immigrant women and non-immigrant Latina women on these measures; 2) To quantify whether there is a correlation between ACTH, cortisol, and PPD and whether there are differences between immigrant and non-immigrant Latina women; 3) To assess the feasibility of enrolling Latinas into a laboratory-based study that includes the collection of venous blood for measurement of oxytocin, ACTH, and cortisol; and 4) Assess the performance of the Spanish language protocol and measures to identify barriers to implementation and address needed modifications prior to large-scale implementation.

Subjects: Sixty prenatal (34 to 37 weeks) Latinas (30 immigrants and 30 U.S.-born) who are between the ages of 18 and 45 will be enrolled. Women with a singleton pregnancy who are Latina, who intend to breastfeed for more than 2 months, who have or do not have a history of depression, and who are willing to be followed for 8 weeks after delivery will be enrolled in the study. Latinas who report maternal or infant disorder that may interfere with breastfeeding; those who endorse substance use, and/or who have or have had a psychiatric disorder (e.g., psychosis or serious personality disorders) other than depression or anxiety will be excluded to minimize risk and confounds with the outcomes of interest.

Methods: There will be four study-time points: prenatal visit, 4- and 12-weeks postpartum phone interviews, and one laboratory visit at 8-weeks postpartum. Participants will be compensating after each interview.

Prenatal Visit: We will collect demographic information; assess depression and anxiety status, as well as breastfeeding intention. During the prenatal visit we will also inquire about acculturation and everyday stressors. English and Spanish validated measures will be used.

Postpartum Phone Interviews: We will inquire about breastfeeding practices and self-efficacy using the Breastfeeding Self-Efficacy-Short Form as well as depression status using the EPDS.

Laboratory Visit: At 8 weeks postpartum, biomarkers will be collected via blood draws during breastfeeding and the cold pressor stress test. Oxytocin will be collected during breastfeeding and adrenocorticotropic hormone (ACTH) and cortisol will be collected after a recovery period and during the cold pressor stress test. Childhood and Border-Crossing Trauma will be collected following the laboratory procedures.

What will be gained: This study will enable us to begin to understand Latinas (immigrant and U.S.-born) neuroendocrine responses to high levels of stress, which will enable us to and determine associations between stress and trauma the development of postpartum depression. This study will also enable us to identify risk factors for postpartum depression among immigrant and U.S.-born Latinas.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal Latina/Hispanic women 34 to 37 weeks
* Latina/Hispanic women 18 and 45 years of age
* Latina/Hispanic women with a singleton pregnancy
* Latina/Hispanic women who intend to breastfeed for more than 2 months
* Latina/Hispanic women who are willing to be followed for 16 weeks

Exclusion Criteria:

* Latina/Hispanic women who report maternal or infant disorder that may interfere with breastfeeding
* Latina/Hispanic women who endorse substance use (alcohol and/or elicit drugs)
* Latina/Hispanic women who have or have had a psychiatric disorder (e.g., psychosis or serious personality disorders) other than depression or anxiety

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Latinas (foreign and U.S.-born)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Postpartum depression | third trimester to 12 weeks postpartum
  Postpartum depression will be assessed using the Edinburgh Postpartum Depression Scale (EPDS), a 10-item questionnaire that helps to identify women who have postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sandraluz Lara-Cinisomo, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States